CLINICAL TRIAL: NCT00133575
Title: ACAM 3000 MVA (Acambis Modified Vaccinia Ankara) Immunization Followed by Dryvax® Vaccination of Healthy Vaccinia-Naïve Adults: A Phase I/II, Placebo-Controlled Study of the Effects of Dose and Route of Administration of MVA on Safety, Reactogenicity and Immunogenicity, Followed by Dryvax® Immunization to Assess Effects of MVA Vaccination on Dryvax® Takes
Brief Title: ACAM 3000 MVA at Harvard Medical School
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05-0010; 5U54AI057159-10 (NIH)
Record Dates: First submitted 2005-08-19; First posted 2005-08-23 (Estimated); Results first posted 2009-07-08 (Estimated); Last update posted 2015-01-05 (Estimated); Status verified 2009-09

CONDITIONS: Smallpox
Keywords: MVA, smallpox, Acambis
MeSH Terms: conditions — Smallpox | interventions — smallpox and monkeypox vaccine modified vaccinia ankara-bavarian nordic

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Group E: ACAM3000 MVA 10^7 ID (Experimental): 10 subjects to receive ACAM3000 MVA dose 10^7 TCID50 via intradermal route on days 0 and 28; 2 subjects to receive placebo via intradermal route on days 0 and 28. Dryvax® smallpox vaccine administered at approximately day 180, dosage 10^8 pfu/ml.
  Interventions: Other: Placebo; Biological: MVA Smallpox Vaccine; Biological: Live vaccinia virus vaccine
- Group F: ACAM3000 MVA 10^8 IM (Experimental): 10 subjects to receive ACAM3000 MVA dose 10^8 TCID50 via intramuscular route on days 0 and 28; 2 subjects to receive placebo via intramuscular route on days 0 and 28. Dryvax® smallpox vaccine administered at approximately day 180, dosage 10^8 pfu/ml.
  Interventions: Biological: MVA Smallpox Vaccine; Biological: Live vaccinia virus vaccine; Other: Placebo
- Group D: ACAM3000 MVA 10^8 SC (Experimental): 10 subjects to receive ACAM3000 MVA dose 10^8 TCID50 via subcutaneous route on days 0 and 28; 2 subjects to receive placebo via subcutaneous route on days 0 and 28. Dryvax® smallpox vaccine administered at approximately day 180, dosage 10^8 pfu/ml.
  Interventions: Biological: MVA Smallpox Vaccine; Other: Placebo; Biological: Live vaccinia virus vaccine
- Group B: ACAM3000 MVA 10^7 IM (Experimental): 10 subjects to receive ACAM3000 MVA dose 10^7 TCID50 via intramuscular route on days 0 and 28; 2 subjects to receive placebo via intramuscular route on days 0 and 28. Dryvax® smallpox vaccine administered at approximately day 180, dosage 10^8 pfu/ml.
  Interventions: Biological: MVA Smallpox Vaccine; Biological: Live vaccinia virus vaccine; Other: Placebo
- Group A: ACAM3000 MVA 10^6 ID (Experimental): 10 subjects to receive ACAM3000 MVA dose 10^6 tissue culture infectious dose 50 (TCID50) via intradermal (ID) route on days 0 and 28; 2 subjects to receive placebo via intradermal route on days 0 and 28. Dryvax® smallpox vaccine administered at approximately day 180, dosage 10^8 pfu/ml.
  Interventions: Other: Placebo; Biological: MVA Smallpox Vaccine; Biological: Live vaccinia virus vaccine
- Group C: ACAM3000 MVA 10^7 SC (Experimental): 10 subjects to receive ACAM3000 MVA dose 10^7 TCID50 via subcutaneous (SC) route on days 0 and 28; 2 subjects to receive placebo via subcutaneous route on days 0 and 28. Dryvax® smallpox vaccine administered at approximately day 180, dosage 10^8 pfu/ml.
  Interventions: Biological: MVA Smallpox Vaccine; Other: Placebo; Biological: Live vaccinia virus vaccine

INTERVENTIONS:
Biological: MVA Smallpox Vaccine — MVA smallpox vaccine (ACAM3000 MVA) administered in two doses approximately 28 days apart in the following dose/route combination: 10^7 or 10^8 TCID50 intramuscularly (IM).
  Arms: Group B: ACAM3000 MVA 10^7 IM; Group F: ACAM3000 MVA 10^8 IM
Biological: MVA Smallpox Vaccine — MVA smallpox vaccine (ACAM3000 MVA) administered in two doses approximately 28 days apart in the following dose/route combination: 10^7 or 10^8 TCID50 subcutaneously (SC).
  Arms: Group C: ACAM3000 MVA 10^7 SC; Group D: ACAM3000 MVA 10^8 SC
Other: Placebo — Sterile saline (0.9%) volume of 0.5 ml intradermally in the deltoid.
  Arms: Group A: ACAM3000 MVA 10^6 ID; Group E: ACAM3000 MVA 10^7 ID
Other: Placebo — Sterile saline (0.9%) volume of 0.5 ml subcutaneously in the deltoid.
  Arms: Group C: ACAM3000 MVA 10^7 SC; Group D: ACAM3000 MVA 10^8 SC
Biological: MVA Smallpox Vaccine — MVA smallpox vaccine (ACAM3000 MVA) administered in two doses approximately 28 days apart in the following dose/route combination: 10^6 or 10^7 TCID50 intradermally (ID).
  Arms: Group A: ACAM3000 MVA 10^6 ID; Group E: ACAM3000 MVA 10^7 ID
Biological: Live vaccinia virus vaccine — Dryvax® smallpox vaccine administered at approximately day 180, dosage 10^8 pfu/ml.
Other: Placebo — Sterile saline (0.9%) volume of 0.5 ml intramuscularly in the deltoid.
  Arms: Group B: ACAM3000 MVA 10^7 IM; Group F: ACAM3000 MVA 10^8 IM

SUMMARY:
The purpose of this study is to assess the safety of an experimental smallpox vaccine (MVA: Modified Vaccinia Ankara) and to compare the body's immune (system that fights disease) response to this vaccine. Participants will be assigned to 1 of 6 study groups. Each group will include 12 subjects, 10 will receive the modified smallpox vaccine and two will receive placebo, an inactive substance. The vaccine will be administered in 1 of 3 ways: under the skin; in the muscle; or between the muscle and the skin. Groups A and B will receive Dryvax® 6-15 months after the initial MVA vaccine; groups C, D, E, and F will receive Dryvax® 6 months after the initial MVA vaccine. Study procedures will include documenting side effects for 14 days after each vaccination, electrocardiogram (picture of the hearts activity) and blood samples. Participants will be involved in study related procedures for up to 18 months.

DETAILED DESCRIPTION:
The emergence of smallpox as a potential agent of bioterrorism has heightened concern about the vulnerability of the population to infection with this agent, and has led to proposals to undertake large scale smallpox immunization of military personnel and "first responders" in the United States, including certain health care workers. A particularly promising vaccine approach to the development of an effective, yet less reactogenic vaccine to smallpox is the use of Modified Vaccinia Ankara (MVA) as a vaccine. Despite the established efficacy of smallpox vaccination, the parameters of protective immunity against smallpox infection are incompletely understood. This is a phase I/II trial to be conducted under a placebo controlled double-blind, randomized allocation of study product. The purpose of this study is to assess the safety and immunogenicity of ACAM 3000 MVA in healthy vaccinia-naïve adult subjects. Participants will include 72 healthy, male or female, from the Boston metropolitan area. Six dose regimens will be studied initially: 10^6 or 10^7 tissue culture infectious dose 50 (TCID50) administered intradermally and 10^7 or 10^8 TCID50 administered intramuscularly or subcutaneously as 2 immunizations 1 month apart. Each arm will be comprised of 12 subjects, 10 of whom will receive ACAM3000 MVA and 2 of whom will receive placebo. A subsequent vaccinia vaccination will be offered to all patients. Consenting participants in Groups A and B will receive the vaccinia (Dryvax®) inoculation between 6 and 15 months after the initial MVA / placebo vaccination. Consenting participants in groups C, D, E and F will receive the Dryvax® inoculation approximately 6 months after the initial MVA / placebo vaccination, coinciding with planned visit 13. Assessment of safety will be carried out by observation and measurement of acute clinical and laboratory evidence of reactions or toxicity; including clinical, electrocardiographic or laboratory evidence of myopericarditis. Assessment of immunogenicity will be carried out by the measurement of humoral and cell-mediated immune response to ACAM 3000 MVA and vaccinia, performed on blood samples obtained at various times prior to and after immunization over the one year period of the study. Response to vaccinia will be assessed clinically (effect on a "take") and the results will be correlated with immune responses to MVA. Subjects will be followed for reactogenicity. Clinical assessments and blood samples will be obtained sequentially for immunogenicity determinations.

ELIGIBILITY:
Inclusion Criteria:

General:

* Age: greater than or equal to 18 and born after 1971.
* Complete a written assessment of understanding prior to enrollment and verbalize understanding of all questions answered incorrectly.
* Informed consent: Be able, willing, and have signed the informed consent form.
* Health: Be in good general health without clinically significant medical history, physical examination findings, or clinically significant abnormal laboratory results. A clinically significant condition or process includes one or more of the following: a) A condition that is chronic or recurring and is life threatening b) A process that would affect the immune response c) A process that would require medication that affects the immune response d) A condition for which repeated injections or blood draws may pose additional risk to the participant e) A condition that requires active medical intervention or monitoring to avert grave danger to the participant's health or well-being f) A condition or process in which signs or symptoms could be confused with reactions to vaccine

Laboratory:

* Willing to have blood samples stored for future smallpox related research.
* Hematology and chemistries within institutional normal limits for age and sex for the following: hemoglobin, white blood cell (WBC)], serum creatinine, platelets, troponin, alanine aminotransferase (ALT) [within 1.25 under normal limits (ULN), aspartate aminotransferase (AST) (within 1.25 ULN), alkaline phos (within 1.25 ULN), total bilirubin (within 1.25 ULN).
* Negative for Hepatitis B surface antigen and Hepatitis C virus (HCV) antibodies [If HCV antibodies are positive, and negative for HCV by polymerase chain reaction (PCR), subject is eligible]
* Negative FDA-approved human immunodeficiency virus (HIV) blood test within 8 weeks prior to enrollment
* Normal urine dipstick or urinalysis:

  1. Negative glucose, and
  2. Negative or trace protein and negative or trace hemoglobin (if trace hemoglobin is present, a urinalysis is required to exclude participants with counts greater than the institutional normal range)

In addition to meeting ALL of the above criteria, FEMALE participants must meet BOTH of the following criteria:

* Negative serum or urine beta-human chorionic gonadotropin (HCG) pregnancy test performed within 24 hours prior to any vaccination.
* Reproductive status: A female participant either must:

  1. not be of reproductive potential. Reproductive potential in women is defined as not having reached menopause (no menses for one year) or having undergone hysterectomy, bilateral oophorectomy, or tubal ligation.
  2. be with a male partner(s) throughout the duration of the study who has undergone successful vasectomy (A vasectomy is considered successful if a woman reports that a male partner has (1) microscopic documentation of azospermia, or (2) a vasectomy more than 2 years ago with no resultant pregnancy despite sexual activity post-vasectomy.), or
  3. agree to avoid pregnancy through alternative methods and agree to consistently use contraception for at least 21 days prior to enrollment until the last protocol visit. Contraception is defined as using one of the following methods:

  i) condoms (male or female with or without a spermicide) ii) diaphragm or cervical cap with spermicide iii) intrauterine device (IUD) iv) hormone-based therapy, e.g., contraceptive pills, Norplant, or Depo-Provera

In addition to the above criteria, female participants must meet the following criteria prior to participating in Dryvax vaccination:

* Negative serum or urine beta-HCG pregnancy test performed within 24 hrs prior to vaccination.
* Comply with one of the following methods of contraception for at least 21 days prior to vaccination and at least 2 months post vaccination.

  1. Hormonal contraception: such as implants, injectables, combined oral contraceptives
  2. Not be of reproductive potential: this may be due to

  i) Hysterectomy or tubal ligation ii) The participant is in a monogamous relationship with a male partner who has undergone successful vasectomy (Successful vasectomy as defined as microscopic documentation of azospermia or a vasectomy more than two years ago with no resultant pregnancy despite sexual activity post-vasectomy.) c) Sexual abstinence

Exclusion Criteria:

* Prior vaccination with a vaccinia product. Determined by clinical evidence of scarification or self-reported history of vaccinia vaccination (such as in the United States military before 1991 or after 2003).
* Immunosuppressive medications within 168 days prior to initial study vaccine administration, e.g., oral/parenteral corticosteroids, and/or cytotoxic medications. Not excluded: A participant using any of the following is not excluded: corticosteroid nasal spray for allergic rhinitis; or topical corticosteroids as prescribed by a physician for an acute, uncomplicated dermatitis; or over the counter medications (including topical corticosteroids for an acute, uncomplicated dermatitis); use of rapidly tapered steroids for an acute isolated condition, which does not include asthma within 28 days prior to vaccine administration.
* Currently using corticosteroid eye drops.
* Receipt of blood products within 120 days prior to initial study vaccine administration.
* Receipt of immunoglobulin within 60 days prior to initial study vaccine administration.
* Receipt of live attenuated vaccines within 30 days prior to initial study vaccine administration.
* Receipt of investigational research agents within 30 days prior to initial study vaccine administration.
* Receipt of medically indicated subunit or killed vaccines, e.g., influenza, pneumococcal, or allergy treatment with antigen injections within 14 days prior to initial study vaccine administration.

Participant has a history of any of the following:

* Acute febrile illness on the day of vaccination.
* Eczema or atopic dermatitis (past or present).
* Chronic exfoliative skin condition.
* Acute skin disorders of large magnitude (greater than 2x2 centimeters), e.g., burns or lacerations.
* History or presence of skin cancer at vaccination site.
* Heart disease including history of a myocardial infarction (MI), angina, congestive heart failure (CHF), or pericardial pathology.
* Ten percent or greater risk of developing a myocardial infarction or coronary death within the next 10 years using the National Cholesterol Education Program's risk assessment tool (http://hin.nhlbi.nih.gov/atpiii/calculator.asp).

NOTE: This criterion applies only to subjects 20 years of age and older AND only if at least one of the following applies:

a) have smoked a cigarette in the past month, and/or b) have hypertension (defined as systolic blood pressure greater than 140 mm Hg) or are on antihypertensive medication, and/or c) have a family history of coronary heart disease in male first-degree relative (father or brother) less than 55 years of age or a female first-degree relative (mother or sister) less than 65 years of age.

* Household contacts/sexual contacts with, or frequent and/or prolonged exposure to any of the following:

  a) Children less than 12 months of age b) Pregnant women or women who are breast feeding c) Individuals with a history of eczema or atopic dermatitis d) Individuals with chronic exfoliative skin disorders or skin disorders of large magnitude (greater than 2x2 centimeters) e) Individuals with an immunosuppressive disorder such as HIV infection, organ transplantation, or a condition requiring prolonged corticosteroid therapy
* Electrocardiogram (ECG) with clinically significant findings, or features that would interfere with the assessment of myo/pericarditis as determined by the consulting cardiologist, including any of the following: (1) Conduction disturbance (complete left or incomplete right bundle branch block or nonspecific intraventricular conduction disturbance with waves of ventricular activity of the heart traced on an ECG (QRS) greater than 120 millisecond (ms), atrioventricular (AV) block of any degree, or QTc prolongation (greater than 440 ms); (2) Repolarization (ST segment or T wave) abnormality; (3) Significant atrial or ventricular arrhythmia; (4) Frequent atrial or ventricular ectopy (e.g. frequent premature atrial contractions, 2 premature ventricular contractions in a row); (5) ST elevation consistent with ischemia; (6) Evidence of past or evolving myocardial infarction.
* Known or suspected allergy to any component of the vaccine or diluent.
* Allergy to eggs or blood products [including immunoglobulin (IgG) or vaccinia immunoglobulin].
* Serious adverse reactions to vaccines including anaphylaxis and related symptoms such as hives, respiratory difficulty, angioedema, and/or abdominal pain. Not excluded: A participant who had an adverse reaction to pertussis vaccine as a child is not excluded.
* Autoimmune disease.
* Immunodeficiency.
* Asthma that is unstable, e.g., use of oral or intravenous corticosteroids, hospitalization or intubation during the past 2 years a) Inhaled steroids are not permissible
* Diabetes mellitus type I or type II including cases controlled with diet alone. Not excluded: A participant with past gestational diabetes is not excluded.
* Bleeding disorder diagnosed by a doctor, e.g., factor deficiency, coagulopathy, or platelet disorder requiring special precautions. Not excluded: A participant who states he/she has easy bruising or bleeding, but does not carry a formal diagnosis and has had intramuscular (IM) injections and blood draws without any adverse experience, is not excluded.
* Seizure disorder not excluded: A participant with a remote history (over 3 years ago) of seizure who has not required medications for over 3 years is not excluded if (a) the seizures were febrile seizures under the age of 2, or (b) secondary to alcohol withdrawal, or (c) if the seizure only occurred once.
* Asplenia. Any condition resulting in the absence or removal of the spleen.
* Psychiatric condition that precludes compliance with the protocol. Specifically excluded are persons with one or more of the following:

  a) Psychoses within the past 5 years. b) Suicidal ideation occurring within 2 years prior to enrollment. Not excluded: A participant with a remote history (greater than 3 years) of a suicide attempt or suicide gesture is not excluded if the investigator finds the participant (a) to be of sound mental health; and (b) the suicide attempt was a well-defined, isolated event; and (c) the cause or inciting factor(s) no longer has relevance to the individual. A participant currently in therapy, due to a suicide attempt or gesture, or suicidal ideation, may be enrolled only when the participant's current therapist or health care provider provides documentation that the participant currently is not suicidal.
* Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence or a participant's ability to give informed consent.
* Female participants: Participant is pregnant and/or breast-feeding.

In addition to the above criteria, the following exclusion criteria apply to those participants consenting to Dryvax vaccination:

-A history of the following:

1. Excessive scarring
2. Known or suspected allergy to any component of the vaccine or diluent including polymyxin B sulfate, dihydrostreptomycin sulfate, chlorotetracycline hydrochloride, neomycin, and phenol.
3. Known allergy to cidofovir or probenecid -Abnormal renal function:

a) A calculated creatinine clearance less than 80 mL/min based on the following formulas: i) Males: [(140 - age in years) X weight in kilograms (kg)]/(72 X serum creatinine) ii) Females: 0.85 X [(140 - age in years) X weight in kg]/(72 X serum creatinine)

Ages: 18 Years to 38 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2005-10; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital - Infectious Diseases, Boston, Massachusetts, United States

REFERENCES:
- [Result] Seaman MS, Wilck MB, Baden LR, Walsh SR, Grandpre LE, Devoy C, Giri A, Noble LC, Kleinjan JA, Stevenson KE, Kim HT, Dolin R. Effect of vaccination with modified vaccinia Ankara (ACAM3000) on subsequent challenge with Dryvax. J Infect Dis. 2010 May 1;201(9):1353-60. doi: 10.1086/651560. PMID 20350190
- [Result] Wilck MB, Seaman MS, Baden LR, Walsh SR, Grandpre LE, Devoy C, Giri A, Kleinjan JA, Noble LC, Stevenson KE, Kim HT, Dolin R. Safety and immunogenicity of modified vaccinia Ankara (ACAM3000): effect of dose and route of administration. J Infect Dis. 2010 May 1;201(9):1361-70. doi: 10.1086/651561. PMID 20350191

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Normal healthy vaccinia-naïve young adults who reside in the greater Boston metropolitan area were recruited for this study between September 29, 2005 and April 23, 2007.
Groups:
- 10^6 TCID50 MVA ID: ACAM3000 Modified Vaccinia Ankara dose 10^6 tissue culture infectious dose 50 (TCID50) via intradermal (ID) route on days 0 and 28
- 10^7 TCID50 MVA IM: ACAM3000 Modified Vaccinia Ankara dose 10^7 tissue culture infectious dose 50 (TCID50) via intramuscular (IM) route on days 0 and 28
- 10^7 TCID50 MVA SC: ACAM3000 Modified Vaccinia Ankara dose 10^7 tissue culture infectious dose 50 (TCID50) via subcutaneous (SC) route on days 0 and 28
- 10^8 TCID50 MVA SC: ACAM3000 Modified Vaccinia Ankara dose 10^8 tissue culture infectious dose 50 (TCID50) via subcutaneous (SC) route on days 0 and 28
- 10^7 TCID50 MVA ID: ACAM3000 Modified Vaccinia Ankara dose 10^7 tissue culture infectious dose 50 (TCID50) via intradermal (ID) route on days 0 and 28
- 10^8 TCID50 MVA IM: ACAM3000 Modified Vaccinia Ankara dose 10^8 tissue culture infectious dose 50 (TCID50) via intramuscular (IM) route on days 0 and 28
- Saline Placebo: Saline placebo via intradermal (ID), intramuscular (IM) or subcutaneous (SC) route at days 0 and 28
Period: Overall Study
Arm/Group | 10^6 TCID50 MVA ID | 10^7 TCID50 MVA IM | 10^7 TCID50 MVA SC | 10^8 TCID50 MVA SC | 10^7 TCID50 MVA ID | 10^8 TCID50 MVA IM | Saline Placebo
Started | 10 | 10 | 10 | 10 | 10 | 10 | 12
Completed | 10 | 10 | 8 | 9 | 6 | 9 | 9
Not Completed | 0 | 0 | 2 | 1 | 4 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10^6 TCID50 MVA ID | 10^7 TCID50 MVA IM | 10^7 TCID50 MVA SC | 10^8 TCID50 MVA SC | 10^7 TCID50 MVA ID | 10^8 TCID50 MVA IM | Saline Placebo | Total
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 12 | 72
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 10 | 10 | 10 | 10 | 12 | 72
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (3.1) | 26.9 (4.7) | 24 (3.9) | 24.7 (4.1) | 26.5 (2.2) | 24.2 (3.6) | 25.6 (3.9) | 25.2 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 5 | 7 | 4 | 8 | 6 | 43
  Male | 3 | 4 | 5 | 3 | 6 | 2 | 6 | 29
Region of Enrollment [Number; unit: participants]
  United States | 10 | 10 | 10 | 10 | 10 | 10 | 12 | 72

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting Moderate or Greater Solicited Local Reactions
Description: Number of participants reporting moderate or greater local reactions solicited on the memory aid as well as by study personnel at follow up visits after either vaccination. Participants are counted only once but may have experienced symptoms on multiple occasions.
Time Frame: 15 days after vaccination
Measure: Number; unit: Participants
Arm/Group | 10^6 TCID50 MVA ID | 10^7 TCID50 MVA IM | 10^7 TCID50 MVA SC | 10^8 TCID50 MVA SC | 10^7 TCID50 MVA ID | 10^8 TCID50 MVA IM | Saline Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 12
Participants
  Erythema | 3 | 0 | 1 | 6 | 9 | 2 | 1
  Induration | 1 | 0 | 1 | 4 | 8 | 2 | 0
  Itchiness at vaccination site | 0 | 0 | 0 | 0 | 2 | 0 | 0
  Limitation of motion | 0 | 0 | 0 | 0 | 0 | 1 | 0
  Pain at injection site | 0 | 0 | 0 | 4 | 1 | 4 | 0
  Tenderness | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Rash | 0 | 2 | 0 | 0 | 1 | 0 | 0

2. Primary Outcome: Number of Participants Reporting Moderate or Greater Solicited Systemic Reactions
Description: Number of participants reporting moderate or greater systemic reactions solicited on the memory aid as well as by study personnel at follow up visits after either vaccination. Participants are counted only once but may have experienced symptoms on multiple occasions.
Time Frame: 15 days after vaccination
Measure: Number; unit: Participants
Arm/Group | 10^6 TCID50 MVA ID | 10^7 TCID50 MVA IM | 10^7 TCID50 MVA SC | 10^8 TCID50 MVA SC | 10^7 TCID50 MVA ID | 10^8 TCID50 MVA IM | Saline Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 12
Participants
  Change in appetite | 1 | 0 | 0 | 0 | 0 | 1 | 0
  Chills | 1 | 1 | 0 | 0 | 0 | 0 | 0
  Feeling tired | 3 | 3 | 0 | 1 | 1 | 4 | 0
  Headache | 1 | 1 | 0 | 0 | 2 | 5 | 0
  Joint pain | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Muscle aches | 2 | 1 | 0 | 2 | 0 | 4 | 0
  Nausea | 0 | 2 | 0 | 0 | 0 | 0 | 0
  Oral temperature elevated | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Underarm pain | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Underarm swelling | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Primary Outcome: Number of Participants With Hematologic Laboratory Abnormalities After Vaccination
Description: Number of participants with hematologic laboratory abnormalities after vaccination, including hemoglobin, white blood cell count, neutrophil count and platelet count. Participants are counted only once for each parameter but may have experienced an abnormality of that parameter on multiple occasions.
Time Frame: 28 days after vaccination
Measure: Number; unit: Participants
Arm/Group | 10^6 TCID50 MVA ID | 10^7 TCID50 MVA IM | 10^7 TCID50 MVA SC | 10^8 TCID50 MVA SC | 10^7 TCID50 MVA ID | 10^8 TCID50 MVA IM | Saline Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 12
Participants
  Hemoglobin | 3 | 2 | 2 | 1 | 2 | 3 | 1
  White blood cells | 4 | 5 | 4 | 2 | 1 | 3 | 5
  Neutrophil count | 3 | 1 | 3 | 0 | 1 | 0 | 1
  Platelets | 1 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Clinical Chemistry Laboratory Abnormalities After Vaccination
Description: Number of participants with clinical chemistry laboratory abnormalities after vaccination, including total bilirubin and serum creatinine. Participants are counted only once for each parameter but may have experienced an abnormality of that parameter on multiple occasions.
Time Frame: 28 days after vaccination
Measure: Number; unit: Participants
Arm/Group | 10^6 TCID50 MVA ID | 10^7 TCID50 MVA IM | 10^7 TCID50 MVA SC | 10^8 TCID50 MVA SC | 10^7 TCID50 MVA ID | 10^8 TCID50 MVA IM | Saline Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 12
Participants
  Bilirubin | 0 | 0 | 2 | 0 | 1 | 1 | 1
  Creatinine | 0 | 0 | 0 | 0 | 0 | 1 | 1

5. Primary Outcome: Number of Participants With Enzymatic Clinical Laboratory Abnormalities After Vaccination
Description: Number of participants with enzymatic clinical laboratory abnormalities after vaccination, including AST, ALT and alkaline phosphatase. Participants are counted only once for each parameter but may have experienced an abnormality of that parameter on multiple occasions
Time Frame: 28 days after vaccination
Measure: Number; unit: Participants
Arm/Group | 10^6 TCID50 MVA ID | 10^7 TCID50 MVA IM | 10^7 TCID50 MVA SC | 10^8 TCID50 MVA SC | 10^7 TCID50 MVA ID | 10^8 TCID50 MVA IM | Saline Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 12
Participants
  AST (SGPT) | 0 | 0 | 0 | 0 | 1 | 0 | 1
  ALT (SGOT) | 0 | 0 | 0 | 0 | 1 | 0 | 0
  Alkaline Phosphatase | 0 | 1 | 0 | 2 | 5 | 1 | 3

6. Primary Outcome: Number of Participants With Urinalysis Laboratory Abnormalies After Vaccination
Description: Number of participants with urinalysis laboratory abnormalies after vaccination, including proteinuria and hematuria by dipstick. Participants are counted only once for each parameter but may have experienced an abnormality of that parameter on multiple occasions.
Time Frame: 28 days after vaccination
Measure: Number; unit: Participants
Arm/Group | 10^6 TCID50 MVA ID | 10^7 TCID50 MVA IM | 10^7 TCID50 MVA SC | 10^8 TCID50 MVA SC | 10^7 TCID50 MVA ID | 10^8 TCID50 MVA IM | Saline Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 12
Participants
  Proteinuria | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Hematuria | 1 | 0 | 0 | 0 | 0 | 0 | 0

7. Primary Outcome: Number of Participants With Signs of Possible Myopericarditis
Description: Number of participants with signs of possible myopericarditis, either by clinical or laboratory (EKG, troponin) evaluation, at any time after vaccination for the during of the study
Time Frame: Within 360 days after vaccination
Measure: Number; unit: Participants
Arm/Group | 10^6 TCID50 MVA ID | 10^7 TCID50 MVA IM | 10^7 TCID50 MVA SC | 10^8 TCID50 MVA SC | 10^7 TCID50 MVA ID | 10^8 TCID50 MVA IM | Saline Placebo
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 12
Participants | 0 | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Peak Neutralizing Antibodies to ACAM3000 MVA
Description: Median neutralizing antibody titers against ACAM3000 MVA as the assay antigen, as assessed from sera collected 2 weeks after receipt of 2 doses.
Time Frame: Approximately Day 42 after first vaccination
Measure: Median (Inter-Quartile Range); unit: Titers
Arm/Group | 10^6 TCID50 MVA ID | 10^7 TCID50 MVA IM | 10^7 TCID50 MVA SC | 10^8 TCID50 MVA SC | 10^7 TCID50 MVA ID | 10^8 TCID50 MVA IM | Saline Placebo
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 10 | 10
Titers | 27 [20 to 76] | 74 [52 to 113] | 68 [51 to 126] | 202 [157 to 569] | 220 [49 to 695] | 333 [177 to 584] | 20 [20 to 20]

9. Secondary Outcome: Peak Neutralizing Antibodies to Vaccinia
Description: Median neutralizing antibody titers against vaccinia virus as the assay antigen, as assessed from sera collected 2 weeks after receipt of 2 doses.
Time Frame: Approximately Day 42 after first vaccination
Measure: Median (Inter-Quartile Range); unit: Titers
Arm/Group | 10^6 TCID50 MVA ID | 10^7 TCID50 MVA IM | 10^7 TCID50 MVA SC | 10^8 TCID50 MVA SC | 10^7 TCID50 MVA ID | 10^8 TCID50 MVA IM | Saline Placebo
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 10 | 10
Titers | 20 [20 to 20] | 20 [20 to 39] | 24 [20 to 32] | 70 [58 to 141] | 129 [41 to 274] | 179 [88 to 237] | 20 [20 to 20]

10. Secondary Outcome: Peak Binding Antibodies (ELISA) to ACAM3000 MVA
Description: Median binding antibody titers against ACAM3000 MVA as the ELISA assay antigen, as assessed from sera collected 2 weeks after receipt of 2 doses.
Time Frame: Approximately Day 42 after first vaccination
Measure: Median (Inter-Quartile Range); unit: Titers
Arm/Group | 10^6 TCID50 MVA ID | 10^7 TCID50 MVA IM | 10^7 TCID50 MVA SC | 10^8 TCID50 MVA SC | 10^7 TCID50 MVA ID | 10^8 TCID50 MVA IM | Saline Placebo
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 10 | 10
Titers | 90 [30 to 810] | 270 [270 to 2430] | 270 [270 to 810] | 810 [810 to 7290] | 2430 [270 to 2430] | 2430 [810 to 2430] | 30 [30 to 30]

11. Secondary Outcome: Peak Binding Antibodies (ELISA) to Vaccinia
Description: Median binding antibody titers against vaccinia virus as the ELISA assay antigen, as assessed from sera collected 2 weeks after receipt of 2 doses.
Time Frame: Approximately Day 42 after first vaccination
Measure: Median (Inter-Quartile Range); unit: Titers
Arm/Group | 10^6 TCID50 MVA ID | 10^7 TCID50 MVA IM | 10^7 TCID50 MVA SC | 10^8 TCID50 MVA SC | 10^7 TCID50 MVA ID | 10^8 TCID50 MVA IM | Saline Placebo
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 10 | 10
Titers | 90 [30 to 270] | 540 [30 to 2430] | 540 [270 to 810] | 4860 [2430 to 7290] | 540 [270 to 2430] | 2430 [810 to 2430] | 30 [30 to 30]

12. Secondary Outcome: Peak T-cell Gamma Interferon Responses (ELISPOT)
Description: Median T-cell gamma interferon responses against the vaccinia virus as the assay antigen, as assessed by ELISPOT from sera collected 2 weeks after receipt of 2 doses. Responses are expressed as the number of spot forming units per 10^6 peripheral blood mononuclear cells (SFU/10^6 PBMC).
Time Frame: Approximately Day 42 after first vaccination
Measure: Median (Inter-Quartile Range); unit: SFU/10^6 PBMC
Arm/Group | 10^6 TCID50 MVA ID | 10^7 TCID50 MVA IM | 10^7 TCID50 MVA SC | 10^8 TCID50 MVA SC | 10^7 TCID50 MVA ID | 10^8 TCID50 MVA IM | Saline Placebo
Number analyzed (Participants) | 10 | 10 | 8 | 10 | 10 | 10 | 10
SFU/10^6 PBMC | 61 [0 to 89] | 373 [175 to 637] | 114 [79 to 279] | 99 [36 to 198] | 38 [14 to 137] | 185 [113 to 377] | 10 [0 to 25]

13. Secondary Outcome: Peak Titer of Viral Shedding Post Dryvax Challenge
Description: Median Dryvax virus titers as assessed from swabs of the vaccination site lesion taken at intervals until the vaccination site is scabbed. The maximum titer recovered during the sampling period for each participant is utilized in determining the median for the group.
Time Frame: Until vaccination site lesion has scabbed
Measure: Median (Full Range); unit: Titers
Arm/Group | 10^6 TCID50 MVA ID | 10^7 TCID50 MVA IM | 10^7 TCID50 MVA SC | 10^8 TCID50 MVA SC | 10^7 TCID50 MVA ID | 10^8 TCID50 MVA IM | Saline Placebo
Number analyzed (Participants) | 2 | 5 | 7 | 6 | 9 | 0 | 7
Titers | 497,000 [99,000 to 895,000] | 52,500 [29,000 to 191,000] | 23,000 [3,150 to 545,000] | 570 [0 to 157,000] | 11,550 [0 to 147,500] |  | 480,000 [32,500 to 2,010,000]

14. Secondary Outcome: Assessment of Dryvax Take Category
Description: Restricted to participants who received Dryvax 6-15 months after MVA. A "take" is a vesicle surrounded by a red areola which becomes umbilicated and then pustular before scabbing. Category 0=No take; Category 1=Significant modified take skin reaction; Category 2=Modified take skin reaction; Category 3=Primary take skin reaction
Time Frame: 3 weeks after Dryvax challenge
Measure: Number; unit: Participants
Arm/Group | 10^6 TCID50 MVA ID | 10^7 TCID50 MVA IM | 10^7 TCID50 MVA SC | 10^8 TCID50 MVA SC | 10^7 TCID50 MVA ID | 10^8 TCID50 MVA IM | Saline Placebo
Number analyzed (Participants) | 2 | 4 | 7 | 6 | 9 | 0 | 7
Participants
  Category 0 | 0 | 0 | 0 | 0 | 0 |  | 0
  Category 1 | 0 | 0 | 0 | 0 | 0 |  | 0
  Category 2 | 0 | 0 | 0 | 0 | 0 |  | 0
  Category 3 | 2 | 4 | 7 | 6 | 9 |  | 7

ADVERSE EVENTS:
Time Frame: Subjects maintained a diary card to record the occurrence of solicited symptoms (vaccine reactogenicity) for 15 days (Day 0-14) after each vaccination. Unsolicited adverse events were collected through Day 360 after the first vaccination.
Description: The solicited symptoms are reported separately after each vaccination. The occurrence of a solicited symptom on any day(s) at any severity within the 15 day period was considered one event.
Arm/Group | 10^6 TCID50 MVA ID | 10^7 TCID50 MVA IM | 10^7 TCID50 MVA SC | 10^8 TCID50 MVA SC | 10^7 TCID50 MVA ID | 10^8 TCID50 MVA IM | Saline Placebo
Serious Adverse Events (participants affected / at risk) | 1/10 | 2/10 | 0/10 | 0/10 | 0/10 | 0/10 | 0/12
Other Adverse Events (participants affected / at risk) | 10/10 | 10/10 | 8/10 | 10/10 | 10/10 | 10/10 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 10^6 TCID50 MVA ID (N=10) | 10^7 TCID50 MVA IM (N=10) | 10^7 TCID50 MVA SC (N=10) | 10^8 TCID50 MVA SC (N=10) | 10^7 TCID50 MVA ID (N=10) | 10^8 TCID50 MVA IM (N=10) | Saline Placebo (N=12)
Amenorrhoea (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | 10^6 TCID50 MVA ID (N=10) | 10^7 TCID50 MVA IM (N=10) | 10^7 TCID50 MVA SC (N=10) | 10^8 TCID50 MVA SC (N=10) | 10^7 TCID50 MVA ID (N=10) | 10^8 TCID50 MVA IM (N=10) | Saline Placebo (N=12)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Visual disturbance (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomach discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site discolouration (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper extremity mass (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Body tinea (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes simplex (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localized infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 6 (9) | 3 (3) | 3 (3) | 3 (3) | 5 (9) | 4 (7) | 4 (4)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pilonidal cyst (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3)
Vaginal candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meniscus lesion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sunburn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood pressure (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure systolic increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram PR prolongation (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart rate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Smear cervix abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lactose intolerance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 4 (4) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope vasovagal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Endodontic procedure (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appetite disorder - post dose 1 (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) — Solicited on the diary card as "Change in appetite"
Appetite disorder - post dose 2 (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0/8 (0) | 0 (0) | 0 (0) | 1 (1) | 0/11 (0) — Solicited on the diary card as "Change in appetite"
Appetite disorder - post Dryvax (Metabolism and nutrition disorders) | 0/2 (0) | 0/5 (0) | 2/7 (2) | 0/6 (0) | 1/9 (1) | 0/0 (0) | 2/7 (2) — Solicited on the diary card as "Change in appetite"
Chills - post dose 1 (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — Solicited on the diary card as "Chills"
Chills - post dose 2 (General disorders) | 2 (2) | 1 (1) | 0/8 (0) | 0 (0) | 0 (0) | 0 (0) | 0/11 (0) — Solicited on the diary card as "Chills"
Chills - post Dryvax (General disorders) | 0/2 (0) | 1/5 (1) | 1/7 (1) | 0/6 (0) | 0/9 (0) | 0/0 (0) | 0/7 (0) — Solicited on the diary card as "Chills"
Injection site erythema - post dose 1 (General disorders) | 7 (7) | 2 (2) | 4 (4) | 6 (6) | 9 (9) | 3 (3) | 3 (3) — Solicited on the diary card as "Erythema (redness)", measured in millimeters
Injection site erythema - post dose 2 (General disorders) | 8 (8) | 1 (1) | 2/8 (2) | 8 (8) | 10 (10) | 4 (4) | 0/11 (0) — Solicited on the diary card as "Erythema (redness)", measured in millimeters
Injection site erythema - post Dryvax (General disorders) | 2/2 (2) | 5/5 (5) | 7/7 (7) | 6/6 (6) | 7/9 (7) | 0/0 (0) | 7/7 (7) — Measured in millimeters at follow up visits by clinic staff
Fatigue - post dose 1 (General disorders) | 3 (3) | 5 (5) | 1 (1) | 4 (4) | 3 (3) | 5 (5) | 1 (1) — Solicited on the diary card as "Feeling tired"
Fatigue - post dose 2 (General disorders) | 3 (3) | 1 (1) | 3/8 (3) | 3 (3) | 3 (3) | 5 (5) | 1/11 (1) — Solicited on the diary card as "Feeling tired"
Fatigue - post Dryvax (General disorders) | 0/2 (0) | 3/5 (3) | 4/7 (4) | 1/6 (1) | 1/9 (1) | 0/0 (0) | 0/7 (0) — Solicited on the diary card as "Feeling tired"
Headache - post dose 1 (Nervous system disorders) | 1 (1) | 4 (4) | 1 (1) | 2 (2) | 5 (5) | 3 (3) | 1 (1) — Solicited on the diary card as "Headache"
Headache - post dose 2 (Nervous system disorders) | 4 (4) | 3 (3) | 1/8 (1) | 0 (0) | 4 (4) | 3 (3) | 0/11 (0) — Solicited on the diary card as "Headache"
Headache - post Dryvax (Nervous system disorders) | 0/2 (0) | 3/5 (3) | 1/7 (1) | 0/6 (0) | 1/9 (1) | 0/0 (0) | 1/7 (1) — Solicited on the diary card as "Headache"
Injection site induration - post dose 1 (General disorders) | 4 (4) | 1 (1) | 2 (2) | 8 (8) | 9 (9) | 1 (1) | 2 (2) — Solicited on the diary card as "Induration (Bump/Swelling)", measured in millimeters
Injection site induration - post dose 2 (General disorders) | 5 (5) | 2 (2) | 2/8 (2) | 8 (8) | 10 (10) | 3 (3) | 0/11 (0) — Solicited on the diary card as "Induration (Bump/Swelling)", measured in millimeters
Injection site induration - post Dryvax (General disorders) | 2/2 (2) | 5/5 (5) | 7/7 (7) | 6/6 (6) | 7/9 (7) | 0/0 (0) | 7/7 (7) — Measured in millimeters at follow up visits by clinic staff
Injection site pruritus - post dose 1 (General disorders) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 6 (6) | 2 (2) | 0 (0) — Solicited on the diary card as "Itchiness at vaccination site"
Injection site pruritus - post dose 2 (General disorders) | 1 (1) | 0 (0) | 2/8 (2) | 6 (6) | 6 (6) | 1 (1) | 0/11 (0) — Solicited on the diary card as "Itchiness at vaccination site"
Injection site pruritus - post Dryvax (General disorders) | 2/2 (2) | 4/5 (4) | 6/7 (6) | 3/6 (3) | 5/9 (5) | 0/0 (0) | 6/7 (6) — Solicited on the diary card as "Itchiness at vaccination site"
Arthralgia - post dose 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) — Solicited on the diary card as "Joint pain"
Arthralgia - post dose 2 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0/8 (0) | 0 (0) | 1 (1) | 0 (0) | 0/11 (0) — Solicited on the diary card as "Joint pain"
Arthralgia - post Dryvax (Musculoskeletal and connective tissue disorders) | 1/2 (1) | 1/5 (1) | 1/7 (1) | 0/6 (0) | 0/9 (0) | 0/0 (0) | 1/7 (1) — Solicited on the diary card as "Joint pain"
Joint range of motion decreased - post dose 1 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) — Solicited on the diary card as "Limitation of motion"
Joint range of motion decreased - post dose 2 (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0/8 (0) | 0 (0) | 0 (0) | 1 (1) | 0/11 (0) — Solicited on the diary card as "Limitation of motion"
Joint range of motion decreased - post Dryvax (Musculoskeletal and connective tissue disorders) | 0/2 (0) | 1/5 (1) | 1/7 (1) | 0/6 (0) | 0/9 (0) | 0/0 (0) | 0/7 (0) — Solicited on the diary card as "Limitation of motion"
Myalgia - post dose 1 (Musculoskeletal and connective tissue disorders) | 1 (1) | 5 (5) | 2 (2) | 3 (3) | 0 (0) | 5 (5) | 1 (1) — Solicited on the diary card as "Muscle aches"
Myalgia - post dose 2 (Musculoskeletal and connective tissue disorders) | 3 (3) | 5 (5) | 1/8 (1) | 0 (0) | 2 (2) | 4 (4) | 0/11 (0) — Solicited on the diary card as "Muscle aches"
Myalgia - post Dryvax (Musculoskeletal and connective tissue disorders) | 1/2 (1) | 2/5 (2) | 3/7 (3) | 0/6 (0) | 0/9 (0) | 0/0 (0) | 2/7 (2) — Solicited on the diary card as "Muscle aches"
Nausea - post dose 1 (Gastrointestinal disorders) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) — Solicited on the diary card as "Nausea"
Nausea - post dose 2 (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0/8 (0) | 2 (2) | 0 (0) | 0 (0) | 0/11 (0) — Solicited on the diary card as "Nausea"
Nausea - post Dryvax (Gastrointestinal disorders) | 0/2 (0) | 0/5 (0) | 2/7 (2) | 0/6 (0) | 1/9 (1) | 0/0 (0) | 1/7 (1) — Solicited on the diary card as "Nausea"
Pyrexia - post dose 1 (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) — Solicited on the diary card as "Temperature", taken orally and considered fever if >= 37.7 degrees celsius
Pyrexia - post dose 2 (General disorders) | 1 (1) | 0 (0) | 0/8 (0) | 0 (0) | 0 (0) | 0 (0) | 0/11 (0) — Solicited on the diary card as "Temperature", taken orally and considered fever if >= 37.7 degrees celsius
Pyrexia - post Dryvax (General disorders) | 0/2 (0) | 0/5 (0) | 1/7 (1) | 0/6 (0) | 0/9 (0) | 0/0 (0) | 0/7 (0) — Solicited on the diary card as "Temperature", taken orally and considered fever if >= 37.7 degrees celsius
Injection site pain - post dose 1 (General disorders) | 2 (2) | 5 (5) | 6 (6) | 8 (8) | 7 (7) | 9 (9) | 1 (1) — Solicited on the diary card as "Pain at injection site"
Injection site pain - post dose 2 (General disorders) | 1 (1) | 5 (5) | 6/8 (6) | 9 (9) | 7 (7) | 6 (6) | 1/11 (1) — Solicited on the diary card as "Pain at injection site"
Injection site pain - post Dryvax (General disorders) | 2/2 (2) | 3/5 (3) | 4/7 (4) | 1/6 (1) | 2/9 (2) | 0/0 (0) | 4/7 (4) — Solicited on the diary card as "Pain at injection site"
Rash - post dose 1 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) — Solicited on the diary card as "Rash"
Rash - post dose 2 (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0/8 (0) | 0 (0) | 0 (0) | 0 (0) | 0/11 (0) — Solicited on the diary card as "Rash"
Tenderness - post dose 1 (General disorders) | 2 (2) | 3 (3) | 2 (2) | 8 (8) | 5 (5) | 0 (0) | 0 (0) — Solicited at follow up visits as "Tenderness"
Tenderness - post dose 2 (General disorders) | 2 (2) | 0 (0) | 3/8 (3) | 4 (4) | 2 (2) | 0 (0) | 1/11 (1) — Solicited at follow up visits as "Tenderness"
Axillary pain - post dose 1 (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) — Solicited on the diary card as "Underarm pain"
Axillary pain - post dose 2 (General disorders) | 0 (0) | 0 (0) | 1/8 (1) | 0 (0) | 0 (0) | 0 (0) | 0/11 (0) — Solicited on the diary card as "Underarm pain"
Axillary pain - post Dryvax (General disorders) | 1/2 (1) | 1/5 (1) | 3/7 (3) | 1/6 (1) | 1/9 (1) | 0/0 (0) | 4/7 (4) — Solicited on the diary card as "Underarm pain"
Swelling - post dose 1 (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Solicited on the diary card as "Underarm swelling"
Swelling - post Dryvax (General disorders) | 0/2 (0) | 1/5 (1) | 1/7 (1) | 1/6 (1) | 1/9 (1) | 0/0 (0) | 4/7 (4) — Solicited on the diary card as "Underarm swelling"

LIMITATIONS AND CAVEATS:
The Dryvax challenge was optional and administered to only a subset of participants before being discontinued prior to being offered to the subjects in the last cohort.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less